CLINICAL TRIAL: NCT04514640
Title: A Quasi-experimental Study Testing a Mindfulness Meditation Mobile App on Sleep and Neurophysiological Outcomes Using the Oura Ring
Brief Title: Calm + Oura Sleep Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Jennifer Huberty, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00012202
Record Dates: First submitted 2020-08-11; First posted 2020-08-17 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Sleep

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General Meditation (Experimental): Participants will be asked to meditate every day during the daytime for at least 10 min/session. Participants can use any general meditation including the "Daily Calm" which can be found on the homepage or by clicking on the "meditate" tab in the app. Participants will be asked to not choose any sleep meditations or Sleep Stories.
  Interventions: Behavioral: The Calm app
- Sleep Meditation (Experimental): Participants will be asked to meditate every day just before going to bed for at least 10 min/session. Participants can use any sleep meditations which can be found by clicking on the "meditate" tab and then "sleep". Particpiants will be asked to not choose any general meditations including the Daily Calm or Sleep Stories.
  Interventions: Behavioral: The Calm app
- Sleep Stories (Experimental): Participants will be asked to listen to a Sleep Story every day just before going to bed for at least 10 min/session. Participants can listen to any Sleep Story which can be found by clicking on the "sleep" tab. Participants will be asked to not choose any general meditations including the Daily Calm or sleep meditations.
  Interventions: Behavioral: The Calm app

INTERVENTIONS:
Behavioral: The Calm app — All participants (n=100) will be asked to download the Calm app to their phone. Participants will then receive an email containing 4-weeks of free access to Calm. All participants be asked to use Calm once per day for at least 10 minutes based on their group assignment (i.e., general meditation during daytime, sleep meditation before bed, or sleep stories before bed). Participants will be asked to turn on the "take a moment" feature in the Oura app in order for the Oura ring to collect neurophysiological measures before, during, and after meditations. Additionally, participants will be asked to complete sleep diaries every day throughout the intervention.

SUMMARY:
This is a quasi-experimental study with pre-post assessment using a convenience sample of Calm and Oura employees. We will employ two weeks of baseline data collection and administer the intervention for four-weeks. Participants will be randomized to one of three groups (i.e., general meditations, sleep meditations, or Sleep Stories). Self-report assessments will be conducted during baseline periods and during week 1 and week 4 of the intervention. Sleep diaries and objective (i.e., Oura ring and Calm app) usage data will be collected on a continual basis during intervention.

The purpose of this study is to:

1. Test the preliminary effects of using Calm (daytime vs nighttime) for four weeks on sleep outcomes (sleep quality, sleep onset, sleep efficiency, number of nighttime awakenings, total sleep time) using self-report and objective measures.

   1. Self-report: Sleep diaries, pre-sleep arousal (Pre-Sleep Arousal Survey), fatigue (Fatigue Severity Scale), daytime sleepiness (Epworth Sleepiness Scale), insomnia (Insomnia Severity Index), sleep quality (Pittsburgh Sleep Quality Index)
   2. Objective: Oura ring (sleep onset, sleep efficiency, number of nighttime awakenings, total sleep time, REM/light/deep sleep).
2. Test the preliminary effects of using Calm (daytime vs nighttime) on neurophysiological outcomes [heart rate variability (HRV), heart rate, respiratory rate] as measured by the Oura ring during meditation and after four-weeks of mobile meditation practice.

DETAILED DESCRIPTION:
More than 30% of the US population reports sleep disturbances, and the Centers for Disease Control and Prevention has identified insufficient sleep as a public health epidemic. Current evidence-based interventions for sleep disturbance (e.g., Cognitive Behavior Therapy for insomnia, Relaxation Therapy) are lengthy and limited due to the need for specialized providers. Pharmaco-therapy may help, however they have inherent limitations (e.g., tolerance, side effects, interactions) to their use. Novel treatments that effectively and conveniently address sleep disturbances (i.e., help individuals self-manage sleep) need further investigation.

Commercially available mobile applications (apps) may help individuals self-manage health conditions conveniently at low cost and with little to no side effects. Specifically, mindfulness-based interventions (e.g., mindfulness meditation) targeting sleep and delivered via a mobile app may be an attractive, feasible and effective solution to improve sleep. Few, if any sleep interventions testing mobile meditation apps have assessed their effects on sleep and most studies only include self-report measures rather than objective measures of sleep (e.g., portable sleep trackers). Additionally, no studies have assessed the neurophysiological changes (heart rate variability, heart rate, respiratory rate) during or with prolonged use of a mindfulness meditation mobile app and whether these changes vary based on time of day. Thus, there is an unexplored opportunity to efficiently and effectively test the use of a mindfulness meditation mobile app on sleep and neurophysiological outcomes.

Findings from our previous study testing the effects of the mindfulness meditation mobile app called Calm on sleep outcomes (manuscript in review; PloS one), suggest that the Calm app improves self-reported sleep quality, and decreases daytime fatigue, daytime sleepiness, and cognitive/somatic pre-sleep arousal in sleep disturbed adults. However, we did not collect any objective data to confirm these findings and are unsure if these findings can be replicated in otherwise healthy adults. We also did not collect any neurophysiological outcomes during meditation practice.

Therefore, the purpose of this study is to:

1. Test the preliminary effects of using Calm (daytime vs nighttime) for four weeks on sleep outcomes (sleep quality, sleep onset, sleep efficiency, number of nighttime awakenings, total sleep time) using self-report and objective measures.

   1. Self-report: Sleep diaries (Pittsburgh Sleep Diaries), pre-sleep arousal (Pre-Sleep Arousal Survey), fatigue (Fatigue Severity Scale), and daytime sleepiness (Epworth Sleepiness Scale), insomnia (Insomnia Severity Index)
   2. Objective: Oura ring (sleep onset, sleep efficiency, number of nighttime awakenings, total sleep time, REM/light/deep sleep).
2. Test the preliminary effects of using Calm (daytime vs nighttime) on neurophysiological outcomes [heart rate variability (HRV), heart rate, respiratory rate] as measured by the Oura ring during meditation and after four-weeks of mobile meditation practice.

The Calm app provides daily, 10-minute, guided general meditations as well as sleep-focused meditations grounded in mindfulness-based stress reduction (MBSR) and Vipassana meditation. Uniquely, Calm also offers "Sleep Stories", developed using techniques from Cognitive Behavioral Therapy and Relaxation Technique.

The Oura Ring is a portable wearable device designed to be worn on the finger. The device includes a 3D accelerometer and gyroscope to measure light, deep, and rapid eye movement sleep. The device also measures heart rate, heart rate variability, and respiratory rate. The Oura Ring has shown promise as a tool to measure sleep outcomes when compared to the gold standard polysomnography.

Study design: This is a quasi-experimental study with pre-post assessment using a convenience sample of Calm and Oura employees. We will employ two weeks of baseline data collection and administer the intervention for four-weeks. Participants will be randomized to one of three groups (i.e., general meditations, sleep meditations, or Sleep Stories). Self-report assessments will be conducted during baseline periods and during week 1 and week 4 of the intervention. Sleep diaries and objective (i.e., Oura ring and Calm app) usage data will be collected on a continual basis during intervention.

ELIGIBILITY:
Inclusion Criteria:

* Employee of Calm or Oura
* >18 years of age
* English speaking
* Willing to download the Calm app to their smartphone
* Willing to wear Oura ring
* Willing to be randomized.

Exclusion Criteria:

* Oura employees who do not own an Oura ring

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Diaries | Daily for 6 weeks
  Sleep diaries assessing sleep/wake time and sleep quality
Pre-Sleep Arousal Survey | Change from baseline pre-sleep arousal at 4-weeks; 16-items (8-items measure cognitive arousal and 8-items measure somatic arousal); Scores range from 8-40 with higher scores indicating greater pre-sleep arousal
  Cognitive and somatic pre-sleep arousal
Fatigue Severity Scale | Change from baseline fatigue at 4-weeks; 9-items; Scores range from 1-7 with higher scores indicating higher levels of fatigue.
  Daytime fatigue
Epworth Sleepiness Scale | Change from baseline daytime sleepiness at 4-weeks; 8-items; Scores range from 0-24 with higher scores indicating higher levels of daytime sleepiness.
  Daytime sleepiness
Insomnia Severity Index | Change from baseline symptoms of insomnia at 4-weeks; 7-items; Scores range from 0-28 with higher scores indicating greater symptoms of insomnia.
  Symptoms of insomnia

SECONDARY OUTCOMES:
Heart rate | Daily for 6 weeks
  beats per minute collected from Oura ring
Heart rate variability | Daily for 6 weeks
  interbeat interval collected from Oura ring
Respiratory rate | Daily for 6 weeks
  Number of breaths per minute collected from Oura ring
Sleep onset | Daily for 6 weeks
  Time went to bed collected from Oura ring
Sleep efficiency | Daily for 6 weeks
  Percent of time in bed compared to total sleep time collected from Oura ring
number of nightime awakenings | Daily for 6 weeks
  Number of times spent awake during the night collected from Oura ring
Total sleep time | Daily for 6 weeks
  Number of minutes slept at night collected from Oura ring
Sleep stages | Daily for 6 weeks
  minutes of sleep spent in rapid eye movement, light, or deep collected from Oura ring

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No